CLINICAL TRIAL: NCT05081830
Title: Suitability, Clinical Utility and Acceptability of an Online Transdiagnostic Intervention for Emotional Disorders and Stress-related Disorders in Mexican Sample: A Randomized Clinical Trial
Brief Title: Online Transdiagnostic Intervention for Emotional Disorders and Stress-related Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Anabel De La Rosa Gomez, PhD, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNAM_FESI_IT300721
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Emotional Disorder; Stress Related Disorder; Anxiety Disorders; Depression
Keywords: online therapy; e-therapy; mexican population; adults; transdiagnostic intervention
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: A randomized controlled study will be carried out, following the guidelines set forth in the CONSORT statement (http://www.consort-statement.org) and CONSORT EHealth ( https://www.jmir.org/2011/4/e126/ ). An experimental design between subjects with three independent groups will be used, with within-subject measurements at four evaluation moments: pretest, posttest, follow-up at 3 and 6 months (Solomon Solomon, Cavanaugh & Draine, 2009). Participants will be randomly assigned to one of three conditions: (a) transdiagnostic intervention via the Internet; (b) Cognitive-Behavior Therapy via the Internet; (c) waiting list control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded: The initial interview by the evaluator will be recorded and the video / audio will be shared with an independent evaluator who does not know the case for evaluation. Once the evaluation is completed, users will be randomly assigned to one of the study conditions. The randomization will be carried out by an independent researcher through the random.stg software in a 1: 1: 1 ratio by saturation of blocks of 12 per condition. The coordinator will inform the participant of the condition in which he / she will participate in the study (experimental or control waiting list) and, depending on the characteristics of said condition, he / she will be discharged from the study and will put him / her in contact with the advisor who has been assigned to you.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transdiagnostic intervention via the Internet (Experimental): Treatment provided in eight individual sessions of 60 min., Once a week by videoconference. The integrity of the treatment will be controlled through the therapist's manual (Barlow et al., 2011) adapted for the Mexican population and to the online modality.
  Interventions: Behavioral: Transdiagnostic online intervention
- TCC intervention via the Internet (Active Comparator): The TCC intervention program is short, with active, focused and directive participation, in 8 individual weekly sessions of one hour by videoconference.
  Interventions: Behavioral: TCC online intervention
- waiting list control. (No Intervention): Participants in the control group on the waiting list will be assigned to the intervention after 2 months after randomization and will join the Transdiagnostic intervention.

INTERVENTIONS:
Behavioral: Transdiagnostic online intervention — Based on the theoretical proposal of Barlow et al. (2011) a treatment applicable to all anxiety and mood disorders (unipolar depression) will be implemented. The unified protocol incorporates proven emotion-focused psychological techniques (Ellard et al., 2010). The main components are: (1) motivation for change, understanding emotions, and recognition and observation of emotional response; (2) learn to observe experiences, evaluate and reevaluate thoughts; (3) what is emotional avoidance, emotion and behavior, and awareness and tolerance of physical sensations; (4) emotional exposure to physical sensations and situations and achievements, maintenance and prevention of relapses.
  Arms: transdiagnostic intervention via the Internet
Behavioral: TCC online intervention — This program incorporates psychological techniques under the cognitive-behavioral model that have demonstrated their effectiveness in online mode (De la Rosa, 2019; Flores et al., 2014). The main components are: (1) psychoeducation, (2) cognitive restructuring, (3) identification and expression of emotions, (4) assertiveness training and (5) problem solving, and (6) relapse prevention. The order of application of each technique is established by the advisor derived from the formulation of treatment of each case to solve the problems raised, under supervision.
  Arms: TCC intervention via the Internet

SUMMARY:
The general objective of this study is to determine the indicators of suitability, clinical utility and satisfaction of the transdiagnostic online intervention for the treatment of emotional disorders and those derived from stress and trauma in a Mexican community sample.

The specific aims are:

* To Carry out a screening evaluation from the transdiagnostic model by evaluating clinical indicators (depression, anxiety, acute / post-traumatic stress, emotional regulation strategies, intolerance to uncertainty) and that allow determining the frequency, intensity and severity of cases identified by type of emotional problem.
* Measure the fidelity of the use of the intervention manual in each treatment condition.
* Evaluate the degree of satisfaction, acceptance, complexity and modality of the transdiagnostic intervention.
* To know the degree of suitability of the transdiagnostic intervention from the point of view of therapists and supervisors in relation to the problems of the studied sample and the recommendations for its improvement.
* To compare the clinical utility of the transdiagnostic intervention via the internet for the treatment of emotional disorders and those derived from stress and trauma against the efficacy of the CBT intervention and the waiting list group.

DETAILED DESCRIPTION:
In recent decades, research findings indicate that cognitive-behavioral interventions, from a disorder-specific perspective, have shown great empirical support and constitute the first-line treatment for anxiety and depression care. However, these treatments are little used. In this regard, various reasons have been noted that explain the limited access and lack of availability to effective interventions; a minority of people actively seek psychological care due to their own condition of emotional distress, for fear of social stigma, for geographical reasons that separate them from health centers, for reasons of time, preference for another type of treatment or self -help, by the high cost of psychological support, which makes it inaccessible and unaffordable for both the user and the public health system. Likewise, it has been exposed that comorbidity between mental disorders, as well as the gap between research findings and clinical practice, could influence the little dissemination of effective treatments; which leads to a lack of up-to-date professionals who provide relevant interventions. Emotional dysregulation of negative affect has been found to be a study factor that is providing relevant data for a better understanding and approach to emotional disorders from a transdiagnostic perspective, a term coined from a dimensional conception to designate effective treatments aimed at two or more specific disorders. Thus, transdiagnostic treatments could help to overcome the drawbacks related to comorbidity between disorders. Now, technological progress has generated alternatives for psychological assistance, both for the evaluation and for the treatment of different emotional disorders. In this regard, the possibilities offered by technologies are highlighted; since the intervention programs supported by the Internet have been empirically tested to achieve effectiveness and efficiency / cost-benefit, and can be key to guaranteeing access to those who the interventions are inaccessible. Thus, the present study has the purpose of knowing the indicators of suitability, clinical utility and satisfaction of the transdiagnostic intervention via videoconferencing for the treatment of emotional disorders and those derived from stress and trauma.

Hypothesis

* The transdiagnostic intervention program via the internet will reduce symptoms of anxiety / depression and / or comorbid acute stress compared to a cognitive-behavioral treatment (CBT) group and a waiting list group.
* The transdiagnosis intervention program via internet will show statistical gains in the reduction of symptoms of anxiety / depression and / or acute stress, and a clinically significant improvement greater than the CBT intervention program and the waiting list group.
* There will be a higher acceptance / satisfaction index reported by the participants in the transdiagnostic intervention program via the internet compared to the CBT intervention and with the group without treatment.
* It will be found that emotional regulation functions as moderating variables of clinical change.
* The changes will be maintained for three and six months after the end of the transdiagnosis intervention program.

ELIGIBILITY:
Inclusion Criteria:

1. be of legal age;
2. voluntarily participate in the study;
3. meet diagnostic criteria for emotional disorders (anxiety or depression) according to the International Neuropsychiatric Interview- Mini, version 5.0, and show a score ≤ 25 on the Beck Anxiety Depression Inventory and / or ≤ 30 on the Inventory Depression of Beck-BDI-II,
4. have access to a computer equipment with an Internet connection, (e) have a valid email address, (f) have basic digital skills in the use of a system operating and internet browsing.

Exclusion Criteria:

1. psychotic disorder;
2. alcohol and drug abuse;
3. medical illness whose severity or characteristics prevent the performance of the intervention;
4. be receiving psychological and / or pharmacological treatment during the study.

Elimination criteria:

1. not accepting the conditions of informed consent
2. absence in two consecutive sessions to the synchronous treatment sessions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrease in the score of Beck Anxiety Inventory | 9 weeks
  Beck Anxiety Inventory ( BAI , Beck & Steer, 1990). Self-applied instrument that consists of 21 questions that determine the severity with which the symptomatic and behavioral categories of anxiety symptoms present in an individual are presented. High internal consistency and adequate construct validity, divergent and convergent (Robles, Varela, Jurado & Páez, 2001).
Decrease in the score of Beck Depression Inventory | 9 weeks
  Beck Depression Inventory (BDI-II; Beck, Steer & Brown, 1996). It consists of 21 items that fundamentally evaluate the clinical symptoms of melancholy and the intrusive thoughts present in depression. Cronbach's alpha for version II (= .87-.92)
Decrease in the score of Checkable List of Post-Traumatic Stress Disorder for DSM-5 (PCL-5) | 9 weeks
  This instrument describes the symptoms of post-traumatic stress taking into consideration the diagnostic criteria of activation, alterations, avoidance and reexperimentation. It has 20 items that are scored on a Likert-type scale that goes from 0 (not at all) to 4 (totally). In its adaptation to the Mexican population, the psychometric properties of the scale show adequate internal consistency with an alpha of .97, as well as an appropriate convergent validity (rs = .58 to .88; Durón-Figueroa et al., 2019).
Decrease in the score of Scale of Difficulties in Emotional Regulation | 9 weeks
  Scale of Difficulties in Emotional Regulation (DERS ; Gratz, & Roemer, 2004). It is a self-applied instrument that measures two dimensions through 15 items, emotional regulation strategies and awareness of emotions. Version validated into Spanish by De la Rosa et al. (2021). Presents Cronbach's alpha between .84-.74.

SECONDARY OUTCOMES:
Increase the level of acceptance and satisfaction of psychological treatment | 9 weeks
  Questionnaire with four questions that report the level of satisfaction with the treatment, if you would recommend the treatment to a friend or relative, is the treatment considered useful for your case and if you think that the treatment was difficult to handle or aversive.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandrina Hernández-Posadas, PhD student, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico; Pablo D Valencia, PhD student, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico; Carolina Santillán-Torres Torija, PhD, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico; Paulina Arenas-Landgrave, PhD, Study Chair — Faculty of Psychology, National Autonomous University of Mexico; Berenice Serrano-Zarate, PhD, Study Chair — Universitat Jaume I; Alejandro Domínguez-Rodríguez, PhD, Study Chair — Valencian International University; Mario F Vázquez-Sánchez, Ms student, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico; Alicia I Flores-Elvira, Ms, Study Chair — Faculty of Higher Studies Iztacala, National Autonomous University of Mexico
Locations (1):
- Faculty of Higher Studies Iztacala, National Autonomous University of Mexico, Tlalnepantla, State of Mexico, Mexico, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a open server of the journal(s) that we will publish the articles that will be the result of this study. The informed consent is already shared in the register of clinical trials.
Supporting Information: Study Protocol, ICF
Time Frame: This data will be available in december 2022 and it will be available for 5 years. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Open access saving personal and sensitive data of the participants.

REFERENCES:
- [Background] Andersson G. Internet-Delivered Psychological Treatments. Annu Rev Clin Psychol. 2016;12:157-79. doi: 10.1146/annurev-clinpsy-021815-093006. Epub 2015 Dec 11. PMID 26652054
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Barlow DH, Allen LB, Choate ML. Toward a Unified Treatment for Emotional Disorders - Republished Article. Behav Ther. 2016 Nov;47(6):838-853. doi: 10.1016/j.beth.2016.11.005. Epub 2016 Nov 10. PMID 27993336
- [Background] Cárdenas, G., Botella, C., Quero, S., De la Rosa, A. & Baños, R. Programa de Telepsicología para el Tratamiento de la Fobia a hablar en público en Población Mexicana. Revista Psicología Iberoamericana. 2014; 22 (1): 45-54.
- [Background] Cárdenas, G., Flores, L. y De la Rosa, A. Psicoterapia vía Internet: Manual de entrenamiento. Facultad de Psicología de la UNAM. DGAPA. 2012. ISBN-978-606-02-2263-4.
- [Background] Ellard KK, Fairholme CP, Boisseau CL, Farchione TJ, Barlow DH. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders: Protocol Development and Initial Outcome Data. Cogn Behav Pract. 2010 Feb;17(1):88-101. doi: 10.1016/j.cbpra.2009.06.002. Epub 2010 Jan 29. PMID 33762811

DOCUMENTS (1):
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05081830/ICF_000.pdf